CLINICAL TRIAL: NCT07374406
Title: A Randomized, Open-label, Single Dose, 2x2 Crossover Study to Evaluate the Safety and Pharmacokinetic Characteristics After Administration of Epaminurad in Healthy Adult Volunteers Under Fasting Conditions
Brief Title: To Evaluate the Safety and Pharmacokinetic Characteristics in Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JW25103
Record Dates: First submitted 2026-01-01; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: randomized, open-label, single dose, 2x2 crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Subjects receive a single dose of Treatment A (JW Pharmaceutical) in Period 1, followed by a washout period, and then a single dose of Treatment B (Shanghai STA Pharmaceutical) in Period 2.
  Interventions: Drug: Epaminurad 9 mg (JW Pharmaceutical); Drug: Epaminurad 9 mg (Shanghai STA Pharmaceutical)
- Group 2 (Experimental): Subjects receive a single dose of Treatment B (Shanghai STA Pharmaceutical) in Period 1, followed by a washout period, and then a single dose of Treatment A (JW Pharmaceutical) in Period 2.
  Interventions: Drug: Epaminurad 9 mg (JW Pharmaceutical); Drug: Epaminurad 9 mg (Shanghai STA Pharmaceutical)

INTERVENTIONS:
Drug: Epaminurad 9 mg (JW Pharmaceutical) — Test product. A single oral dose of 1 tablet containing 9 mg of Epaminurad.
Drug: Epaminurad 9 mg (Shanghai STA Pharmaceutical) — Reference product. A single oral dose of 1 tablet containing 9 mg of Epaminurad.

SUMMARY:
A randomized, open-label, single dose, 2x2 crossover study to evaluate the safety and pharmacokinetic characteristics after administration of Epaminurad in healthy adult volunteers under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

1. Age: 19~55
2. Weight: at least 50 kg for males and 45 kg for females. Body Mass Index(BMI): 18.0 kg/m^2 or heavier and below 30.0 kg/m^2

Exclusion Criteria:

1. Medical history- chronic liver disease, acute gout attack, uric acid stone, diabetes, hypertension, hyperlipidemia or lipid abnormality
2. Clinical examination- eGFR (CKD-EPI) < 60mL/min/1.73m^2, AST (SGOT), ALT (SGPT) > upper limit of normal ranges X 2, CK > upper limit of normal ranges X 5, Positive serologic results Cystatin C > 1.26mg/L

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-01-14 (Actual); Primary Completion 2026-04-19 (Estimated); Study Completion 2026-04-19 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | 3 days
  To evaluate the AUC of Epaminurad
Peak plasma concentrations (Cmax) | 3 days
  To evaluate the Cmax of Epaminurad

CONTACTS AND LOCATIONS:
Overall Officials: Seol Ju Moon, Principal Investigator — Jeonbuk National University Hospital
Locations (1):
- Jeonbuk National University Hospital, Jeonju, South Korea

IPD SHARING:
Plan to Share IPD: No